CLINICAL TRIAL: NCT03643380
Title: Acute Study to Evaluate a Novel Implantable Midfield Powered Device in Humans With Urinary Incontinence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuspera Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: NSM-001
Record Dates: First submitted 2018-07-13; First posted 2018-08-22 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Investigational SNS device (Experimental)
  Interventions: Device: AHLeveeS System

INTERVENTIONS:
Device: AHLeveeS System — AHLeveeS System for treatment of overactive bladder

SUMMARY:
A pre-market, prospective, non-randomized acute feasibility study for the treatment of patients with urinary incontinence (UI) as a consequence of urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

* Subject was eligible for treatment and indication for the Medtronic InterStim system or InterStim II
* Subject wished to undergo an InterStim or InterStim II implant procedure after this acute clinical investigation
* Subject was in good health in the opinion of the investigator
* Subject was able to understand and voluntarily signed and dated the Ethics Committee approved informed consent form prior to initiation of any screening or study-specific procedures
* Subject was minimum of 18 years and maximum of 65 years of age

Exclusion Criteria:

- Subject had any of the contraindications for the InterStim system or InterStim II system

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2018-01-30 (Actual)

PRIMARY OUTCOMES:
Sacral Nerve Response measured by observed bellow response and big toe flexion | Procedure
  Stimulation of the S3 sacral nerve measured by observed bellows response and big toe flexion
AHLeveeS System placement in the S3 foramen assessed by fluoroscopy image | Procedure
  Confirm that the AHLeveeS System can be correctly placed and inserted in close proximity of the sacral nerve in the S3 foramina assessed by fluoroscopy image

CONTACTS AND LOCATIONS:
Overall Officials: Gommert A. van Koeveringe, Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No